CLINICAL TRIAL: NCT01449019
Title: The Contribution of Glucagon-like Peptide 1 (GLP-1) to the Entero-insulinar Axis in Healthy Subjects and Patients With Type 2 Diabetes Mellitus (T2DM)
Brief Title: The Role of Endogenous Glucagon-like Peptide 1 (GLP-1) in Type 2 Diabetes Mellitus (T2DM)
Acronym: DFG_5
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Joerg Schirra, Principal investigator, Clinical Professor, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DPI
Record Dates: First submitted 2011-10-02; First posted 2011-10-07 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GLP-1; Exendin(9-39); Insulin; Glucagon; T2DM; incretin effect; human physiology
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — exendin (9-39); Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intravenous infusion (Active Comparator)
  Interventions: Drug: exendin(9-39)amide; Drug: saline
- intraduodenal perfusion (Experimental)
  Interventions: Other: duodenal meal; Other: duodenal saline

INTERVENTIONS:
Drug: exendin(9-39)amide — intravenous infusion of exendin(9-39)
  Arms: intravenous infusion
Drug: saline — intravenous infusion of saline
  Arms: intravenous infusion
Other: duodenal meal — duodenal perfusion of a meal
  Arms: intraduodenal perfusion
Other: duodenal saline — duodenal perfusion of saline
  Arms: intraduodenal perfusion

SUMMARY:
The purpose of the study is to determine the contribution of endogenous Glucagon-like peptide 1 (GLP-1) to the postprandial secretion of insulin and glucagon and the incretin effect in healthy subjects and patients with type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* male or female (postmenopausal, surgically sterile or using double-barrier method of contraception) healthy subjects and patients with type 2 diabetes mellitus (T2DM)
* must be able to complete a 1 week wash-out of current anti-diabetic medications
* Age 30-70 years
* HbA1c (Hemoglobin A1c) ≤11% at screening
* Body mass index (BMI) <40 kg/m2
* Patients with type 2 diabetes mellitus (T2DM): Must have a fasting blood glucose of ≤12.2 mmol/L (240 mg/dL) at screening
* Able to provide written informed consent prior to study participation
* Able to communicate well with the investigator and comply with the requirements of the study

Exclusion Criteria:

* Patients with type 1 diabetes mellitus (T1DM), diabetes as a result of pancreatic injury, or secondary forms of diabetes (eg Cushing, acromegaly)
* Need for insulin within the previous 3 months
* Use of Thiazolidinediones in the previous 4 weeks
* Significant concomitant disease or complications of diabetes (i.e. nephropathy, autonomic dysfunction, orthostasis).
* Treatment with systemic steroids and thyroid hormone (unstable dosage).
* Patients with any history of gastrointestinal surgery, e.g. partial bowel resections, partial gastric resections, etc.
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing.
* Significant illness within the two weeks prior to dosing.
* Past medical history of clinically significant ECG abnormalities or a family history of a prolonged QT-interval syndrome.
* History of clinically significant drug allergy; history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to the study drug or drugs similar to the study drug.
* history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection;
* history or clinical evidence of pancreatic injury or pancreatitis;
* history or presence of impaired renal function as indicated by abnormal creatinine or urea val-ues or abnormal urinary constituents (e.g., albuminuria);
* evidence of urinary obstruction or difficulty in voiding at screening;
* Polymorphonuclears <1500/µL at inclusion or platelet count < 100,000/μL at screening and baseline.
* History of immunocompromise.
* Evidence of liver disease as indicated by abnormal transaminases and alkaline phosphatase exceeding twice the upper limit of the normal range, and serum bilirubin should not exceed the value of 27 µmol/L (1.6 mg/dL).

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-12; Primary Completion 2007-08 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The incretin effect | Area Under Curve (AUC) Time Frame: from 0 to 90 minutes under duodenal meal perfusion
  The incretin effect is the difference between postprandial plasma concentrations of insulin and C-peptide, respectively, and those during the isoglycemic fasting control experiment. The AUC is calculated after priming intravenous infusion (saline or exendin(9-39)) and under steady state duodenal meal perfusion.

SECONDARY OUTCOMES:
Plasma concentrations of glucagon | Area Under Curve (AUC) Time Frame: from 0 to 90 minutes under duodenal meal perfusion
  The AUC is calculated after priming intravenous infusion (saline or exendin(9-39)) and under steady state duodenal meal perfusion.
Plasma concentrations of insulin | Area Under Curve (AUC) Time Frame: from 0 to 90 minutes under duodenal meal perfusion
  The AUC is calculated after priming intravenous infusion (saline or exendin(9-39)) and under steady state duodenal meal perfusion.
Plasma concentrations of C-peptide | Area Under Curve (AUC) Time Frame: from 0 to 90 minutes under duodenal meal perfusion
  The AUC is calculated after priming intravenous infusion (saline or exendin(9-39)) and under steady state duodenal meal perfusion.
Plasma concentrations of Glucagon-like peptide-1(7-36) (GLP-1(7-36)) | Area Under Curve (AUC) Time Frame: from 0 to 90 minutes under duodenal meal perfusion
  The AUC is calculated after priming intravenous infusion (saline or exendin(9-39)) and under steady state duodenal meal perfusion.
Plasma concentrations of Glucose-dependent insulinotropic polpypeptide (GIP) | Area Under Curve (AUC) Time Frame: from 0 to 90 minutes under duodenal meal perfusion
  The AUC is calculated after priming intravenous infusion (saline or exendin(9-39)) and under steady state duodenal meal perfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Schirra, MD, Principal Investigator — Clinical Research Unit (CRU), Department of Internal Medicine, Campus Großhadern, Clinical Center of Ludwig-Maximilians-University of Munich
Locations (2):
- Germany (2):
  - Ludwig Maximilians-University, Clinical Research Unit, Munich
  - Clinical Research unit, Dept. of Internal Medicine II - Großhadern, University of Munich, Munich

REFERENCES:
- [Derived] Woerle HJ, Carneiro L, Derani A, Goke B, Schirra J. The role of endogenous incretin secretion as amplifier of glucose-stimulated insulin secretion in healthy subjects and patients with type 2 diabetes. Diabetes. 2012 Sep;61(9):2349-58. doi: 10.2337/db11-1701. Epub 2012 Jun 20. PMID 22721966